CLINICAL TRIAL: NCT01451437
Title: A Phase I Study to Evaluate the Safety and Tolerability and Pharmacokinetic/Pharmacodynamics of MK-8242 Administered Alone and in Combination With Chemotherapy in Subjects With Refractory or Recurrent Acute Myelogenous Leukemia (Protocol No. P07649 (005))
Brief Title: Study of MK-8242 Alone and in Combination With Cytarabine in Participants With Acute Myelogenous Leukemia (P07649)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07649; 2011-000709-31 (EudraCT Number); MK-8242-005 (Other: Merck study number)
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Acute Myelogenous Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Pt 1 Arm A: MK-8242 30 mg QD (Experimental): Participants received MK-8242 30 mg once daily (QD) monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 60 mg QD (Experimental): Participants received MK-8242 60 mg QD monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 120 mg QD (Experimental): Participants received MK-8242 120 mg QD monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 250 mg QD (Experimental): Participants received MK-8242 250 mg QD monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 120 mg BID (Experimental): Participants received MK-8242 120 mg twice daily (BID) monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles (except Cycle 1 Day 7 on which MK-8242 120 mg was administered QD in the morning) in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 170 mg BID (Experimental): Participants received MK-8242 170 mg BID monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles (except Cycle 1 Day 7 on which MK-8242 170 mg was administered QD in the morning) in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 210 mg BID (Experimental): Participants received MK-8242 210 mg BID monotherapy on Days 1-7 of a 21-day cycle up to a maximum of 12 cycles (except Cycle 1 Day 7 on which MK-8242 210 mg was administered QD in the morning) in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 250 mg BID (Experimental): Participants received MK-8242 250 mg BID monotherapy on Days 1-7 and Days 15-21 of a 28-day cycle up to a maximum of 12 cycles (except Cycle 1 Day 7 on which MK-8242 250 mg was administered QD in the morning) in Part 1 Arm A.
  Interventions: Drug: MK-8242
- Pt 1 Arm A: MK-8242 300 mg BID (Experimental): Participants received MK-8242 300 mg BID monotherapy on Days 1-7 of a 21-day cycle up to a maximum of 12 cycles (except Cycle 1 Day 7 on which MK-8242 300 mg was administered QD in the morning) in Part 1 Arm A.
  Interventions: Drug: MK-8242

INTERVENTIONS:
Drug: MK-8242 — MK-8242 capsules, orally, once per day on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7) up to a maximum of 12 cycles. Starting dose will be 30 mg and will be escalated in successive cohorts until maximum tolerated dose (MTD) is established. Beginning at a dose level of ≥120 mg total daily dose (TDD), the dosing regimen will switch to twice daily (BID). Amendment 4 added a 21-day dosing cycle in which MK-8242 would be given BID on Days 1-7 of each cycle, at the assigned dose level.
  Other Names: SCH 900242

SUMMARY:
This is a study of MK-8242 alone and in combination with cytarabine in adult participants with refractory or recurrent acute myelogenous leukemia (AML). The study will have 2 Arms. Arm A is for participants with refractory or recurrent AML who are considered ineligible for standard chemotherapy. In Part 1 of Arm A, participants will receive MK-8242 monotherapy in escalating doses to determine the recommended phase 2 dose [RP2D]. In Part 2, participants will receive monotherapy with MK-8242 to confirm the RP2D and assess preliminary efficacy. Arm B is for participants with recurrent AML following an initial complete remission (CR) or CR with incomplete marrow recovery (CRi) of 6 to 12 months duration. In Part 1 of Arm B, participants will receive MK-8242 in escalating doses + cytarabine to determine the RP2D in combination with cytarabine. In Part 2, participants will receive MK-8242 + cytarabine to confirm the RP2D and assess preliminary efficacy. The pharmacokinetics of MK-8242 will be studied in both arms. With Amendment 4 (22 August 2013) a 21-day dosing cycle is added, with MK-8242 being given on Days 1-7 of each 21-day cycle in both the monotherapy and combination therapy arms; data from Arm A will be used to determine whether a participant receives 21-day or 28-day therapy in Arm B.

ELIGIBILITY:
Inclusion criteria:

* For Arm A Part 1 (monotherapy/dose escalation): refractory or recurrent AML, not an appropriate candidate for standard therapy
* For Arm A Part 2 (monotherapy/dose confirmation/cohort expansion): refractory or recurrent AML, not an appropriate candidate for standard therapy, and have wild type p53 gene mutation analysis
* For Arm B Part 1 (combination therapy/dose escalation): recurrent AML having achieved an initial CR or CRi of 6-12 months duration and age ≥18 years old and <70 years old
* For Arm B Part 2 (combination therapy/dose confirmation/cohort expansion): recurrent AML having achieved an initial CR or CRi of 6-12 months duration, age ≥18 years old and <70 years old, and have wild type P53 gene mutation analysis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 for all Arm A, or 0 or 1 for all Arm B
* Negative pregnancy test within 72 hours of the first dose of study medication
* Female participants and male participants and their partners who are of childbearing potential must agree to abstain from sexual intercourse or to use an acceptable method of contraception during the study and for 90 days following the last dose of study therapy
* Adequate organ function
* Recovered from the effects of any prior surgery, radiotherapy or anti-neoplastic treatment, with the exception of alopecia
* Must be able to swallow, retain, and absorb oral medications and oral nutrition
* Must follow the appropriate washout period for prohibited treatments

Exclusion criteria:

* Active malignancy other than AML
* Leptomeningeal leukemia requiring intrathecal therapy
* For Arm A and B, Part 1 only: history of myelodysplastic syndrome (MDS)
* For Arm A and B, Part 2: AML in the background of MDS may be included
* Isolated extramedullary leukemia without also meeting bone marrow criteria for acute leukemia
* AML blast crisis of chronic myelogenous leukemia (CML)
* Bone marrow transplant with active graft-versus host disease (GVHD) or who receives immunosuppressive therapy
* Uncontrolled active infection that requires systemic treatment
* Clinically significant hepatitis at Screening, or hepatitis C antibody positive, hepatitis B surface antigen positive, or human immunodeficiency virus (HIV) seropositive
* Persistent, unresolved, drug-related toxicity
* Breast-feeding, pregnant, intends to become pregnant or intends to breast feed during the study or has a positive pregnancy test at Screening
* A person participating in any other clinical study with a potentially therapeutic agent or who has received another investigational product within 5 half-lives (if the half-life is known) or 28 days (if the half-life is unknown) prior to Day 1 of cycle 1
* A participant who, within the past 6 months, has had any of the following: myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack, or uncontrolled seizure disorder (i.e., seizures within the past 6 months)
* A participant who, at the time of Screening, presents with: unstable or uncontrolled angina, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality
* Known bleeding disorder, e.g. hemophilia or disseminated intravascular coagulopathy or on anti-coagulation therapy
* For Arm B only: Known hypersensitivity to cytarabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2014-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ravandi F, Gojo I, Patnaik MM, Minden MD, Kantarjian H, Johnson-Levonas AO, Fancourt C, Lam R, Jones MB, Knox CD, Rose S, Patel PS, Tibes R. A phase I trial of the human double minute 2 inhibitor (MK-8242) in patients with refractory/recurrent acute myelogenous leukemia (AML). Leuk Res. 2016 Sep;48:92-100. doi: 10.1016/j.leukres.2016.07.004. Epub 2016 Jul 25. PMID 27544076
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=P07649&kw=P07649&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participant in Part 1 received combination therapy (MK-8242 + cytarabine). Study Part 2 was not performed due to early termination of the study.
Groups:
- Pt 1 Arm A: MK-8242 30 mg QD: Participants received MK-8242 30 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 60 mg QD: Participants received MK-8242 60 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 120 mg QD: Participants received MK-8242 120 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 250 mg QD: Participants received MK-8242 250 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 120 mg BID: Participants received MK-8242 120 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 120 mg was administered QD in the morning) in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 170 mg BID: Participants received MK-8242 170 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 170 mg was administered QD in the morning) in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 210 mg BID: Participants received MK-8242 210 mg BID monotherapy on Days 1-7 of each 21-day cycle (except Cycle 1 Day 7 on which MK-8242 210 mg was administered QD in the morning) in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 250 mg BID: Participants received MK-8242 250 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 250 mg was administered QD in the morning) in Part 1 Arm A.
- Pt 1 Arm A: MK-8242 300 mg BID: Participants received MK-8242 300 mg BID monotherapy on Days 1-7 of each 21-day cycle (except Cycle 1 Day 7 on which MK-8242 300 mg was administered QD in the morning) in Part 1 Arm A.
Period: Overall Study
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Started | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Physician Decision | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 1 | 1 | 3 | 2 | 3 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID | Total
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (NA) — not calculated for n=1 | 74.0 (NA) — not calculated for n=1 | 72.3 (6.7) | 77.0 (NA) — not calculated for n=1 | 58.8 (18.5) | 63.3 (14.6) | 63.5 (11.5) | 72.3 (12.5) | 41.0 (14.3) | 62.2 (15.5)
Age, Customized [Number; unit: Participants]
  Adults between 18 and 64 years | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 4 | 12
  From 65 to 84 years | 0 | 1 | 3 | 1 | 2 | 2 | 3 | 2 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 6
  Male | 1 | 1 | 2 | 1 | 4 | 2 | 3 | 3 | 3 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 1 | 1 | 3 | 1 | 4 | 3 | 5 | 3 | 3 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic Or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic Or Latino | 1 | 1 | 3 | 1 | 3 | 2 | 5 | 3 | 3 | 22
  Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were identified using Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0 for toxicities attributable to the study drug. Hematologic DLTs were defined in the absence of morphological evidence of acute leukemia in the marrow if 1) bone marrow: aplastic marrow with <5% cellularity without erythroid, myeloid, or megakaryocytic precursors and 2) peripheral blood: absolute neutrophil count (ANC) <100/µL, platelet count <10,000/µL, and transfusion-dependent anemia. Non-hematologic DLTs were defined as any ≥Grade 3 toxicity with the following exceptions/clarifications: 1) infection, fatigue, anorexia, or alopecia are not included in determination of the DLT 2) Grade 3 nausea, vomiting, diarrhea, or dehydration occurring in a setting of inadequate treatment 3) any abnormal non-hematological laboratory value ≥Grade 3 will be considered a DLT after 72 hours of appropriate medical intervention if not related to an underlying disease or not attributable to another event.
Time Frame: Up to 28 days (Cycle 1) for non-hematologic toxicities and 42 days (Cycle 1) for hematologic toxicities
Population: DLT-evaluable Population: participants who received at least one dose of MK-8242 and completed Cycle 1 of Part 1 or discontinued due to reason of toxicity.
Measure: Number; unit: Participants
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Complete Remission (CR) at RP2D
Description: Clinical activity of MK-8242 given as monotherapy in participants with refractory or recurrent AML measured as participants who achieved CR according to Cheson (2003) criteria at the RP2D. The outcome analysis was not performed since the RP2D for MK-8242 monotherapy could not be established due to early termination of the study.
Time Frame: End of Treatment (up to 198 days)
Population: Full Analysis Set for Efficacy: all participants with confirmed p53 wild type (WT) status who received at least one dose of MK-8242 and have at least one baseline and one post-baseline efficacy assessment.
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Complete Remission With Incomplete Marrow Recovery (CRi) at RP2D
Description: Clinical activity of MK-8242 given as monotherapy in participants with refractory or recurrent AML measured as participants who achieved CRi according to Cheson (2003) criteria at the RP2D. The outcome analysis was not performed since the RP2D for MK-8242 monotherapy could not be established due to early termination of the study.
Time Frame: End of Treatment (up to 198 days)
Population: Full Analysis Set for Efficacy: all participants with confirmed p53 WT status who received at least one dose of MK-8242 and have at least one baseline and one post-baseline efficacy assessment.
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With CR at Dose Levels Other Than RP2D
Description: Clinical activity of MK-8242 given as monotherapy in participants with refractory or recurrent AML measured as participants who achieved CR according to Cheson (2003) criteria at dose levels other than RP2D. CR is defined as a morphologic leukemia-free state with a neutrophil count ≥1,000/µL, a platelet count ≥100,000/µL, no extramedullary disease, and RBC transfusion independence. Presented outcome values are not stratified for dose levels other than RP2D; the RP2D for MK-8242 monotherapy could not be established due to early termination of the study.
Time Frame: End of Treatment (up to 198 days)
Population: Modified Full Analysis Set for Efficacy: all participants with confirmed p53 WT status who received at least one dose of MK-8242.
Measure: Number; unit: Participants
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With CRi at Dose Levels Other Than RP2D
Description: Clinical activity of MK-8242 given as monotherapy in participants with refractory or recurrent AML measured as participants who achieved CRi according to Cheson (2003) criteria at dose levels other than RP2D. CRi is defined as fulfillment of all CR criteria with exceptions for residual neutropenia (<1,000/µL), thrombocytopenia (<100,000/µL), and RBC transfusion dependence. Presented outcome values are not stratified for dose levels other than RP2D; the RP2D for MK-8242 monotherapy could not be established due to early termination of the study.
Time Frame: End of Treatment (up to 198 days)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 6 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24hr) for MK-8242 Alone and in Combination With Cytarabine
Description: AUC(0-24hr) defined as AUC from time zero to 24 hours was determined for Cycle 1 Days 1 and 7 of MK-8242 QD and BID dosing using the trapezoidal up/log trapezoidal down method. For the BID arms, a projection beyond the last sampled time was made if a linear terminal elimination phase half-life was identified with three time-points after Tmax. Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: Cycle 1, Day 1 and Day 7 (QD arms: predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, and 24 hrs postdose; BID arms: predose and 0.5, 1, 2, 4, 6, 8, 12 [optional], and 24 [Day 7 only] hrs postdose)
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (AUC0-24hr) at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 5 | 3 | 3
hr*nM
  Day 1 (n=1,1,3,1,3,2,4,3,1) | 604 (NA) — n/a: not calculated for n=1 | 510 (NA) — n/a: not calculated for n=1 | 3710 (126) | 10900 (NA) — n/a: not calculated for n=1 | 3230 (101) | 6940 (127.0) | 6400 (76.4) | 7910 (81.5) | 9480 (NA) — n/a: not calculated for n=1
  Day 7 (n=1,1,3,1,3,3,5,3,3) | 665 (NA) — n/a: not calculated for n=1 | 515 (NA) — n/a: not calculated for n=1 | 3460 (54.6) | 6840 (NA) — n/a: not calculated for n=1 | 4180 (41.2) | 8440 (105) | 11200 (53.0) | 8800 (56.9) | 14200 (62.5)

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Last (AUC0-last) for MK-8242 Alone and in Combination With Cytarabine
Description: AUC(0-last) defined as AUC from time zero to the time of last quantifiable sample was determined for Cycle 1 Days 1 and 7 of MK-8242 QD and BID dosing using the trapezoidal up/log trapezoidal down method. Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: Cycle 1, Day 1 and Day 7 (QD arms: predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 24, and 48 [Day 7 only] hrs postdose; BID arms: predose and 0.5, 1, 2, 4, 6, 8, 12 [optional], 24 [Day 7 only], 48 [Day 7 only] hrs postdose)
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (AUC0-last) at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 5 | 3 | 3
hr*nM
  Day 1 | 323 (NA) — n/a: not calculated for n=1 | 482 (NA) — n/a: not calculated for n=1 | 3420 (156) | 10900 (NA) — n/a: not calculated for n=1 | 2710 (58.3) | 4370 (111) | 5310 (56.1) | 6710 (76.3) | 7200 (15.1)
  Day 7 | 470 (NA) — n/a: not calculated for n=1 | 482 (NA) — n/a: not calculated for n=1 | 3180 (73.5) | 6830 (NA) — n/a: not calculated for n=1 | 3100 (73.1) | 9560 (183) | 11900 (59.8) | 9080 (51.4) | 15200 (74.1)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) for MK-8242 Alone and in Combination With Cytarabine
Description: AUC0-∞ defined as AUC from time zero to infinity was determined for Cycle 1 Day 7 of MK-8242 QD and BID dosing using the trapezoidal up/log trapezoidal down method. Projection beyond the last sampled time was made if a linear terminal elimination phase half-life was identified with three time-points after Tmax (condition not met for 60 QD and 120 BID dose groups). Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: Cycle 1 Day 7 (QD arms: predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 24, and 48 hrs postdose; BID arms: predose and 0.5, 1, 2, 4, 6, 8, 12 [optional], 24, 48 hrs postdose)
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (AUC0-∞) at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 2 | 2
hr*nM | 650 (NA) — n/a: not calculated for n=1 |  | 3570 (61.6) | 6990 (NA) — n/a: not calculated for n=1 |  | 6480 (NA) — n/a: not calculated for n=1 | 13300 (84.2) | 11700 (40.3) | 15100 (112.0)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-8242 Alone and in Combination With Cytarabine
Description: Cmax was determined for Cycle 1 Days 1 and 7 of MK-8226 QD and BID dosing. Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: as for outcome 7
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (Cmax) at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 5 | 3 | 3
nM
  Day 1 (n=1,1,3,1,4,3,5,3,3) | 56.7 (NA) — n/a: not calculated for n=1 | 109 (NA) — n/a: not calculated for n=1 | 416 (81.4) | 1270 (NA) — n/a: not calculated for n=1 | 561 (51.9) | 984 (93.2) | 1310 (52.5) | 1510 (65.7) | 1940 (25.8)
  Day 7 (n=1,1,3,1,3,3,5,3,3) | 88.8 (NA) — n/a: not calculated for n=1 | 178 (NA) — n/a: not calculated for n=1 | 530 (55.9) | 1320 (NA) — n/a: not calculated for n=1 | 744 (56.1) | 1200 (65.2) | 1550 (50.7) | 1500 (108) | 1920 (80.8)

10. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8242 Alone and in Combination With Cytarabine
Description: Tmax was determined for Cycle 1 Days 1 and 7 of MK-8226 QD and BID dosing. Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: as for outcome 7
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (Tmax) at the time of assessment.
Measure: Median (Full Range); unit: Hours
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 4 | 3 | 5 | 3 | 3
Hours
  Day 1 (n=1,1,3,1,4,3,5,3,3) | 6.25 [NA to NA] — n/a: not calculated for n=1 | 2.00 [NA to NA] — n/a: not calculated for n=1 | 4.00 [2.08 to 4.05] | 4.00 [NA to NA] — n/a: not calculated for n=1 | 4.00 [2.12 to 4.00] | 2.00 [2.00 to 4.13] | 2.00 [1.87 to 4.08] | 2.00 [2.00 to 4.00] | 2.08 [2.00 to 6.00]
  Day 7 (n=1,1,3,1,3,3,5,3,3) | 2.00 [NA to NA] — n/a: not calculated for n=1 | 2.00 [NA to NA] — n/a: not calculated for n=1 | 2.00 [1.00 to 2.00] | 2.00 [NA to NA] — n/a: not calculated for n=1 | 4.00 [2.00 to 4.00] | 4.15 [2.25 to 6.00] | 4.00 [2.00 to 6.00] | 2.00 [1.92 to 4.08] | 4.00 [4.00 to 6.00]

11. Secondary Outcome: Apparent Terminal Half-life (t1/2) for MK-8242 Alone and in Combination With Cytarabine
Description: Elimination phase t1/2 was determined for Cycle 1 Day 7 of MK-8242 QD and BID dosing. Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: as for outcome 8
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (at least three time-points after Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 2 | 2
hr | 4.7 (NA) — n/a: not calculated for n=1 |  | 5.33 (23.5) | 4.57 (NA) — n/a: not calculated for n=1 |  | 10.30 (NA) — n/a: not calculated for n=1 | 7.92 (31.6) | 5.21 (17.9) | 7.06 (36.6)

12. Secondary Outcome: Accumulation Ratio (R) of MK-8242 Alone and in Combination With Cytarabine
Description: The accumulation ratio (R) at steady state (based on dosing interval and apparent terminal half-life (t1/2)) for MK-8242 alone was not determined due to confounding of results by significant concentrations of a drug metabolite (M16). Analysis for the combination therapy was not performed due to early termination of the study (Study Arm B was not performed).
Time Frame: Cycle 1 Day 7 (QD arms: predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 24, and 48 hrs postdose; BID arms: predose and 0.5, 1, 2, 4, 6, 8, 12 [optional], 24 [Day 7 only], 48 [Day 7 only] hrs postdose)
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (R) at the time of assessment.
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Urine Concentration of MK-8242 (Part 2 Arm A Only)
Description: The urine concentration of MK-8242 assessed as a measure of drug bioavailability was not determined due to early termination of the study (Study Part 2 was not performed).
Time Frame: Day 1 (predose and postdose) and Day 7 (postdose)
Population: Participants who received at least one dose of MK-8242, were compliant with study procedures, and had available pharmacokinetic data (urine concentration) at the time of assessment
Groups:
- Pt 2 Arm A: MK-8242 30 mg QD: Participants to receive MK-8242 30 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 60 mg QD: Participants to receive MK-8242 60 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 120 mg QD: Participants to receive MK-8242 120 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 250 mg QD: Participants to receive MK-8242 250 mg QD monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 120 mg BID: Participants to receive MK-8242 120 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 120 mg to be administered QD in the morning) in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 170 mg BID: Participants to receive MK-8242 170 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 170 mg to be administered QD in the morning) in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 210 mg BID: Participants to receive MK-8242 210 mg BID monotherapy on Days 1-7 of each 21-day cycle (except Cycle 1 Day 7 on which MK-8242 210 mg to be administered QD in the morning) in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 250 mg BID: Participants to receive MK-8242 250 mg BID monotherapy on Days 1-7 and Days 15-21 of each 28-day cycle (except Cycle 1 Day 7 on which MK-8242 250 mg to be administered QD in the morning) in Part 2 Arm A.
- Pt 2 Arm A: MK-8242 300 mg BID: Participants to receive MK-8242 300 mg BID monotherapy on Days 1-7 of each 21-day cycle (except Cycle 1 Day 7 on which MK-8242 300 mg to be administered QD in the morning) in Part 2 Arm A.
Arm/Group | Pt 2 Arm A: MK-8242 30 mg QD | Pt 2 Arm A: MK-8242 60 mg QD | Pt 2 Arm A: MK-8242 120 mg QD | Pt 2 Arm A: MK-8242 250 mg QD | Pt 2 Arm A: MK-8242 120 mg BID | Pt 2 Arm A: MK-8242 170 mg BID | Pt 2 Arm A: MK-8242 210 mg BID | Pt 2 Arm A: MK-8242 250 mg BID | Pt 2 Arm A: MK-8242 300 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 7.6 months
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Arm/Group | Pt 1 Arm A: MK-8242 30 mg QD | Pt 1 Arm A: MK-8242 60 mg QD | Pt 1 Arm A: MK-8242 120 mg QD | Pt 1 Arm A: MK-8242 250 mg QD | Pt 1 Arm A: MK-8242 120 mg BID | Pt 1 Arm A: MK-8242 170 mg BID | Pt 1 Arm A: MK-8242 210 mg BID | Pt 1 Arm A: MK-8242 250 mg BID | Pt 1 Arm A: MK-8242 300 mg BID
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 2/3 | 1/1 | 1/4 | 1/3 | 5/6 | 3/3 | 2/4
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 1/1 | 4/4 | 3/3 | 6/6 | 3/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt 1 Arm A: MK-8242 30 mg QD (N=1) | Pt 1 Arm A: MK-8242 60 mg QD (N=1) | Pt 1 Arm A: MK-8242 120 mg QD (N=3) | Pt 1 Arm A: MK-8242 250 mg QD (N=1) | Pt 1 Arm A: MK-8242 120 mg BID (N=4) | Pt 1 Arm A: MK-8242 170 mg BID (N=3) | Pt 1 Arm A: MK-8242 210 mg BID (N=6) | Pt 1 Arm A: MK-8242 250 mg BID (N=3) | Pt 1 Arm A: MK-8242 300 mg BID (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt 1 Arm A: MK-8242 30 mg QD (N=1) | Pt 1 Arm A: MK-8242 60 mg QD (N=1) | Pt 1 Arm A: MK-8242 120 mg QD (N=3) | Pt 1 Arm A: MK-8242 250 mg QD (N=1) | Pt 1 Arm A: MK-8242 120 mg BID (N=4) | Pt 1 Arm A: MK-8242 170 mg BID (N=3) | Pt 1 Arm A: MK-8242 210 mg BID (N=6) | Pt 1 Arm A: MK-8242 250 mg BID (N=3) | Pt 1 Arm A: MK-8242 300 mg BID (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 2 (6) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (4) | 4 (4) | 2 (2) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 1 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the Sponsor. The Investigator further agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.